CLINICAL TRIAL: NCT04165967
Title: A Phase I Study of Adoptive Tumor-infiltrating Lymphocyte Transfer in Combination With Nivolumab in Patients With Advanced Melanoma
Brief Title: Adoptive Tumor-infiltrating Lymphocyte Transfer With Nivolumab for Melanoma
Acronym: BaseTIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: GMP network of Basel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01908; me18Laeubli
Record Dates: First submitted 2019-11-05; First posted 2019-11-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-08

CONDITIONS: Advanced Melanoma
Keywords: Tumor-infiltrating Lymphocyte (TIL) Transfer; Nivolumab; metastatic melanoma; anti-PD-1 therapy; failed immunotherapy; personalized Investigational Medicinal Product (IMP)
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: Tumor-infiltrating infiltrate will be expanded from resected melanoma samples from the patient and expanded TILs will be transferred to the patient after non-myeloablative chemotherapy with cyclophosphamide and fludarabine. TIL transfer will be combined with low dose IL-2 and nivolumab anti-PD-1 treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-infiltrating lymphocyte product (TIL) transfer (Experimental): The TIL product will be produced from excised tumor lesions from the patient. Expanded TILs will be transferred to the patient after non-myeloablative chemotherapy with cyclophosphamide and fludarabine. TIL transfer will be combined with low dose IL-2 and nivolumab anti-PD-1 treatment. The transplant product will be produced in the Good Manufacturing Practice (GMP) facility of the University Hospital in Basel. TIL transfer to Patient at Day 0.
  Interventions: Drug: Combination of TIL Transfer with anti-PD-1 Therapy and low dose IL-2

INTERVENTIONS:
Drug: Combination of TIL Transfer with anti-PD-1 Therapy and low dose IL-2 — The study uses a personalized IMP, i.e. TIL product and in combination with IL-2 treatment and nivolumab.
  Day 0: Autologous TIL: (minimum 5 x 109 and up to a maximum of 2 x 1011 lymphocytes) administered intravenously over 20 to 30 minutes.
  Day 0: Interleukin-2 (Proleukin): 125.000 IU/kg/day s.c. for maximum 12 days as inpatients with a 2 days break after the first 4-5 doses (maximum 10 days dosing). Actual body weight will be used in calculating the dose of interleukin-2.
  Starting Day 14: Nivolumab application 240 mg i.v. over 30 minutes ever 2 weeks with a maximum to 2 years, or until disease progression or inacceptable toxicity.
  Other Names: TIL Transfer; anti-PD-1 Therapy Nivolumab; low dose IL-2

SUMMARY:
This study is to investigate safety and feasibility of a combination therapy of a tumor infiltrating lymphocytes (TIL) transfer with anti-programmed cell death protein (PD)-1 therapy in patients with metastatic melanoma that failed immunotherapy.Tumor-infiltrating lymphocytes will be expanded from resected melanoma samples from the patient and expanded TILs will be transferred to the patient after non-myeloablative chemotherapy with cyclophosphamide and fludarabine. TIL transfer will be combined with low dose Interleukin (IL)-2 and nivolumab anti-PD-1 treatment.

The study uses a personalized Investigational Medicinal Product (IMP), i.e. TIL product and in combination with IL-2 treatment and nivolumab.

DETAILED DESCRIPTION:
Adoptive cell therapy has been previously shown to be an effective treatment option for patients with melanoma. Due to an immunosuppressive microenvironment, not all patients respond to this therapy. In this trial, the immune suppressive microenvironment will be targeted by adding a PD-1 blocking antibody in combination with a TIL Transfer. Tumor-infiltrating lymphocytes will be expanded from resected melanoma samples from the patient and expanded TILs will be transferred to the patient after non-myeloablative chemotherapy with cyclophosphamide and fludarabine. TIL transfer will be combined with low dose IL-2 and nivolumab anti-PD-1 treatment. The study uses a personalized IMP, i.e. TIL product and in combination with IL-2 treatment and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or metastatic melanoma
* At least 1 PD-1 targeted immunotherapy and BRAF inhibition in case of BRAF mutated melanoma
* Resectable tumor mass and measurable disease by CT or MRI per RECIST 1.1 criteria (in addition to the resected lesion)
* World Health Organization (WHO) clinical performance Status (ECOG) 0-1
* Adequate organ function
* Patients of both genders must be willing to practice a highly effective method of birth control during treatment and for five months after receiving the last dose of nivolumab for women and seven months for men
* Patients must be able to understand and sign the Informed consent document
* Hematology: Absolute neutrophil count greater than 1.5 x 109/L without support of filgrastim. Platelet count greater than 100 x 109/L. Hemoglobin greater than 5 mmol/L, or 80 g/L.
* Chemistry: Serum alanine aminotransferase (ALAT)/ aspartate transaminase (ASAT) less than 3 times the upper limit of normal, unless patients have liver metastases (< 5 times ULN). Serum creatinine clearance 50 ml/min or higher. Total Bilirubin less than or equal to 20 micromol/L, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 50 micromol/L. Lactate dehydrogenase (LDH) ≤ 2x ULN
* Serology: Seronegative for HIV antibody. Seronegative for hepatitis B antigen, and hepatitis C antibody. Seronegative for syphilis.

Exclusion Criteria:

* Life expectancy of less than three months
* Patients with metastatic ocular/ mucosal or other non-cutaneous melanoma.
* Requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within the last 3 weeks prior to randomization
* Uncontrolled central nervous system (CNS) metastases. Controlled CNS metastases must be for at least 4 weeks stable.
* Documented Forced expiratory volume at one second (FEV1) less than or equal to 50% predicted for patients with:
* A prolonged history of cigarette smoking (greater than 20 pack/year within the past 2 years)
* Symptoms of respiratory distress
* All patients' toxicities due to prior non-systemic treatment must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures or focal palliative radiotherapy (to non-target lesions) within the past 4 weeks, as long as all toxicities have recovered to grade 1 or less.
* Women who are pregnant or breastfeeding, because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Any active systemic infections, coagulation disorders or other active major medical illnesses.
* Contraindication for IL-2 or nivolumab (allergies etc.).
* Any autoimmune disease: patients with a documented history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, autoimmune thyroiditis (e.g. Hashimoto's disease), autoimmune hepatitis, systemic progressive sclerosis (scleroderma), Systemic Lupus Erythematosus, autoimmune vasculitis (e.g., Wegener's Granulomatosis). Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barré Syndrome) are excluded from this study. Patients with vitiligo are eligible to enter the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | First 3 months during treatment
  Number of Adverse Events to analyze safety of the combination of TIL transfer with IL-2 therapy
Change in body temperature (Degree Celsius) | at each treatment visit (Day 0, and for maximum 12 days as inpatients with a 2 days break after the first 4-5 doses (maximum 10 days dosing)
  Change in Vital signs ( body temperature) to analyze the safety of the combination of TIL transfer with IL-2 therapy
Change in blood pressure (mmHg) | at each treatment visit (Day 0, and for maximum 12 days as inpatients with a 2 days break after the first 4-5 doses (maximum 10 days dosing)
  Change in Vital signs ( blood pressure) to analyze the safety of the combination of TIL transfer with IL-2 therapy
Change in heart beat (beats/minute) | at each treatment visit (Day 0, and for maximum 12 days as inpatients with a 2 days break after the first 4-5 doses (maximum 10 days dosing)
  Change in Vital signs (heart beat) to analyze the safety of the combination of TIL transfer with IL-2 therapy
Change in respiratory frequency (inspiration/minute) | at each treatment visit (Day 0, and for maximum 12 days as inpatients with a 2 days break after the first 4-5 doses (maximum 10 days dosing)
  Change in Vital signs (respiratory frequency) to analyze the safety of the combination of TIL transfer with IL-2 therapy
Change in full blood Counts (number of cells) | at each treatment visit (every 2 weeks) from Day 0= Baseline to week 42
  Change in Laboratory Parameter (full blood counts) to analyze haematological toxicity

SECONDARY OUTCOMES:
Overall Response Rate (ORR) fluorodeoxyglucose (FDG)-positron emission tomography (PET)/CT scan | First 3 months after TIL administration
  Changes of Tumor volume according to RECIST 1.1
Progression Free Survival (PFS) | between pre-treatment and 3-months post-treatment
  Progression free survival, defined as the time between registration to progression or death whichever occurs first.
Overall Survival (OS) defined as the time between registration to death due to any cause | 2 years after TIL transfer
  Overall survival will be measured from the beginning of the treatment to the death of the patient or to survival status analysis acquired during the last follow up.
Tumor response according to revised Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | between pre-treatment and 3-months post-treatment
  Tumor response according to revised Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Objective response rate (ORR) | 2 years after TIL transfer
  In order to assess the objective response rate CT scans and FDG-PET/CT scans will be performed. Response will be measured by best reduction of tumor volume according to RECIST 1.1
Number of Adverse Events according to CTCAE 4.0 | 2 years after TIL transfer
  Overall Safety during whole treatment period analyzed by collection of Adverse Events according to CTCAE 4.0
Metabolic Response | during the first 3 months after TIL transfer
  Response measured by 18FDG-uptake
Number of Serious Adverse Events according to CTCAE 4.0 | 2 years after TIL transfer
  Overall Safety during whole treatment period analyzed by collection of Serious Adverse Events according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Läubli, Prof., Principal Investigator — Division of Medical Oncology and Cancer Immunology, University Hospital Basel; Alfred Zippelius, Prof., Study Chair — Division of Medical Oncology and Cancer Immunology, University Hospital Basel
Locations (1):
- Division of Medical Oncology and Cancer Immunology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Schadendorf D, van Akkooi ACJ, Berking C, Griewank KG, Gutzmer R, Hauschild A, Stang A, Roesch A, Ugurel S. Melanoma. Lancet. 2018 Sep 15;392(10151):971-984. doi: 10.1016/S0140-6736(18)31559-9. PMID 30238891
- [Background] Grob JJ, Garbe C, Ascierto P, Larkin J, Dummer R, Schadendorf D. Adjuvant melanoma therapy with new drugs: should physicians continue to focus on metastatic disease or use it earlier in primary melanoma? Lancet Oncol. 2018 Dec;19(12):e720-e725. doi: 10.1016/S1470-2045(18)30596-5. PMID 30507438
- [Background] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao CD, Wagstaff J, Schadendorf D, Ferrucci PF, Smylie M, Dummer R, Hill A, Hogg D, Haanen J, Carlino MS, Bechter O, Maio M, Marquez-Rodas I, Guidoboni M, McArthur G, Lebbe C, Ascierto PA, Long GV, Cebon J, Sosman J, Postow MA, Callahan MK, Walker D, Rollin L, Bhore R, Hodi FS, Larkin J. Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2017 Oct 5;377(14):1345-1356. doi: 10.1056/NEJMoa1709684. Epub 2017 Sep 11. PMID 28889792
- [Background] Rosenberg SA. Karnofsky Memorial Lecture. The immunotherapy and gene therapy of cancer. J Clin Oncol. 1992 Feb;10(2):180-99. doi: 10.1200/JCO.1992.10.2.180. No abstract available. PMID 1732421
- [Background] Rosenberg SA. Progress in human tumour immunology and immunotherapy. Nature. 2001 May 17;411(6835):380-4. doi: 10.1038/35077246. PMID 11357146
- [Background] Rosenberg SA, Yannelli JR, Yang JC, Topalian SL, Schwartzentruber DJ, Weber JS, Parkinson DR, Seipp CA, Einhorn JH, White DE. Treatment of patients with metastatic melanoma with autologous tumor-infiltrating lymphocytes and interleukin 2. J Natl Cancer Inst. 1994 Aug 3;86(15):1159-66. doi: 10.1093/jnci/86.15.1159. PMID 8028037
- [Background] Rosenberg SA, Spiess P, Lafreniere R. A new approach to the adoptive immunotherapy of cancer with tumor-infiltrating lymphocytes. Science. 1986 Sep 19;233(4770):1318-21. doi: 10.1126/science.3489291.
- [Background] Mills CD, North RJ. Expression of passively transferred immunity against an established tumor depends on generation of cytolytic T cells in recipient. Inhibition by suppressor T cells. J Exp Med. 1983 May 1;157(5):1448-60. doi: 10.1084/jem.157.5.1448. PMID 6189937
- [Background] Fernandez-Cruz E, Woda BA, Feldman JD. Elimination of syngeneic sarcomas in rats by a subset of T lymphocytes. J Exp Med. 1980 Oct 1;152(4):823-41. doi: 10.1084/jem.152.4.823. PMID 6968337
- [Background] Greenberg PD, Kern DE, Cheever MA. Therapy of disseminated murine leukemia with cyclophosphamide and immune Lyt-1+,2- T cells. Tumor eradication does not require participation of cytotoxic T cells. J Exp Med. 1985 May 1;161(5):1122-34. doi: 10.1084/jem.161.5.1122. PMID 3921652
- [Background] Eberlein TJ, Rosenstein M, Rosenberg SA. Regression of a disseminated syngeneic solid tumor by systemic transfer of lymphoid cells expanded in interleukin 2. J Exp Med. 1982 Aug 1;156(2):385-97. doi: 10.1084/jem.156.2.385. PMID 6980254
- [Background] Overwijk WW, Theoret MR, Finkelstein SE, Surman DR, de Jong LA, Vyth-Dreese FA, Dellemijn TA, Antony PA, Spiess PJ, Palmer DC, Heimann DM, Klebanoff CA, Yu Z, Hwang LN, Feigenbaum L, Kruisbeek AM, Rosenberg SA, Restifo NP. Tumor regression and autoimmunity after reversal of a functionally tolerant state of self-reactive CD8+ T cells. J Exp Med. 2003 Aug 18;198(4):569-80. doi: 10.1084/jem.20030590. PMID 12925674
- [Background] Antony PA, Piccirillo CA, Akpinarli A, Finkelstein SE, Speiss PJ, Surman DR, Palmer DC, Chan CC, Klebanoff CA, Overwijk WW, Rosenberg SA, Restifo NP. CD8+ T cell immunity against a tumor/self-antigen is augmented by CD4+ T helper cells and hindered by naturally occurring T regulatory cells. J Immunol. 2005 Mar 1;174(5):2591-601. doi: 10.4049/jimmunol.174.5.2591. PMID 15728465
- [Background] Rooney CM, Smith CA, Ng CY, Loftin S, Li C, Krance RA, Brenner MK, Heslop HE. Use of gene-modified virus-specific T lymphocytes to control Epstein-Barr-virus-related lymphoproliferation. Lancet. 1995 Jan 7;345(8941):9-13. doi: 10.1016/s0140-6736(95)91150-2. PMID 7799740
- [Background] Walter EA, Greenberg PD, Gilbert MJ, Finch RJ, Watanabe KS, Thomas ED, Riddell SR. Reconstitution of cellular immunity against cytomegalovirus in recipients of allogeneic bone marrow by transfer of T-cell clones from the donor. N Engl J Med. 1995 Oct 19;333(16):1038-44. doi: 10.1056/NEJM199510193331603. PMID 7675046
- [Background] Dudley ME, Wunderlich JR, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry RM, Marincola FM, Leitman SF, Seipp CA, Rogers-Freezer L, Morton KE, Nahvi A, Mavroukakis SA, White DE, Rosenberg SA. A phase I study of nonmyeloablative chemotherapy and adoptive transfer of autologous tumor antigen-specific T lymphocytes in patients with metastatic melanoma. J Immunother. 2002 May-Jun;25(3):243-51. doi: 10.1097/01.CJI.0000016820.36510.89. PMID 12000866
- [Background] Rosenberg SA, Aebersold P, Cornetta K, Kasid A, Morgan RA, Moen R, Karson EM, Lotze MT, Yang JC, Topalian SL, et al. Gene transfer into humans--immunotherapy of patients with advanced melanoma, using tumor-infiltrating lymphocytes modified by retroviral gene transduction. N Engl J Med. 1990 Aug 30;323(9):570-8. doi: 10.1056/NEJM199008303230904. PMID 2381442
- [Background] Shahinian VB, Muirhead N, Jevnikar AM, Leckie SH, Khakhar AK, Luke PP, Rizkalla KS, Hollomby DJ, House AA. Epstein-Barr virus seronegativity is a risk factor for late-onset posttransplant lymphoroliferative disorder in adult renal allograft recipients. Transplantation. 2003 Mar 27;75(6):851-6. doi: 10.1097/01.TP.0000055098.96022.F7. PMID 12660514
- [Background] Curtis RE, Travis LB, Rowlings PA, Socie G, Kingma DW, Banks PM, Jaffe ES, Sale GE, Horowitz MM, Witherspoon RP, Shriner DA, Weisdorf DJ, Kolb HJ, Sullivan KM, Sobocinski KA, Gale RP, Hoover RN, Fraumeni JF Jr, Deeg HJ. Risk of lymphoproliferative disorders after bone marrow transplantation: a multi-institutional study. Blood. 1999 Oct 1;94(7):2208-16. PMID 10498590
- [Background] Dudley ME, Gross CA, Langhan MM, Garcia MR, Sherry RM, Yang JC, Phan GQ, Kammula US, Hughes MS, Citrin DE, Restifo NP, Wunderlich JR, Prieto PA, Hong JJ, Langan RC, Zlott DA, Morton KE, White DE, Laurencot CM, Rosenberg SA. CD8+ enriched "young" tumor infiltrating lymphocytes can mediate regression of metastatic melanoma. Clin Cancer Res. 2010 Dec 15;16(24):6122-31. doi: 10.1158/1078-0432.CCR-10-1297. Epub 2010 Jul 28. PMID 20668005
- [Background] Besser MJ, Shapira-Frommer R, Treves AJ, Zippel D, Itzhaki O, Hershkovitz L, Levy D, Kubi A, Hovav E, Chermoshniuk N, Shalmon B, Hardan I, Catane R, Markel G, Apter S, Ben-Nun A, Kuchuk I, Shimoni A, Nagler A, Schachter J. Clinical responses in a phase II study using adoptive transfer of short-term cultured tumor infiltration lymphocytes in metastatic melanoma patients. Clin Cancer Res. 2010 May 1;16(9):2646-55. doi: 10.1158/1078-0432.CCR-10-0041. Epub 2010 Apr 20. PMID 20406835
- [Background] Donia M, Junker N, Ellebaek E, Andersen MH, Straten PT, Svane IM. Characterization and comparison of 'standard' and 'young' tumour-infiltrating lymphocytes for adoptive cell therapy at a Danish translational research institution. Scand J Immunol. 2012 Feb;75(2):157-67. doi: 10.1111/j.1365-3083.2011.02640.x. PMID 21955245
- [Background] Radvanyi LG, Bernatchez C, Zhang M, Fox PS, Miller P, Chacon J, Wu R, Lizee G, Mahoney S, Alvarado G, Glass M, Johnson VE, McMannis JD, Shpall E, Prieto V, Papadopoulos N, Kim K, Homsi J, Bedikian A, Hwu WJ, Patel S, Ross MI, Lee JE, Gershenwald JE, Lucci A, Royal R, Cormier JN, Davies MA, Mansaray R, Fulbright OJ, Toth C, Ramachandran R, Wardell S, Gonzalez A, Hwu P. Specific lymphocyte subsets predict response to adoptive cell therapy using expanded autologous tumor-infiltrating lymphocytes in metastatic melanoma patients. Clin Cancer Res. 2012 Dec 15;18(24):6758-70. doi: 10.1158/1078-0432.CCR-12-1177. Epub 2012 Oct 2. PMID 23032743
- [Background] Andersen RS, Thrue CA, Junker N, Lyngaa R, Donia M, Ellebaek E, Svane IM, Schumacher TN, Thor Straten P, Hadrup SR. Dissection of T-cell antigen specificity in human melanoma. Cancer Res. 2012 Apr 1;72(7):1642-50. doi: 10.1158/0008-5472.CAN-11-2614. Epub 2012 Feb 6. PMID 22311675
- [Background] Kvistborg P, Shu CJ, Heemskerk B, Fankhauser M, Thrue CA, Toebes M, van Rooij N, Linnemann C, van Buuren MM, Urbanus JH, Beltman JB, Thor Straten P, Li YF, Robbins PF, Besser MJ, Schachter J, Kenter GG, Dudley ME, Rosenberg SA, Haanen JB, Hadrup SR, Schumacher TN. TIL therapy broadens the tumor-reactive CD8(+) T cell compartment in melanoma patients. Oncoimmunology. 2012 Jul 1;1(4):409-418. doi: 10.4161/onci.18851. PMID 22754759
- [Background] Robbins PF, Lu YC, El-Gamil M, Li YF, Gross C, Gartner J, Lin JC, Teer JK, Cliften P, Tycksen E, Samuels Y, Rosenberg SA. Mining exomic sequencing data to identify mutated antigens recognized by adoptively transferred tumor-reactive T cells. Nat Med. 2013 Jun;19(6):747-52. doi: 10.1038/nm.3161. Epub 2013 May 5. PMID 23644516
- [Background] van Rooij N, van Buuren MM, Philips D, Velds A, Toebes M, Heemskerk B, van Dijk LJ, Behjati S, Hilkmann H, El Atmioui D, Nieuwland M, Stratton MR, Kerkhoven RM, Kesmir C, Haanen JB, Kvistborg P, Schumacher TN. Tumor exome analysis reveals neoantigen-specific T-cell reactivity in an ipilimumab-responsive melanoma. J Clin Oncol. 2013 Nov 10;31(32):e439-42. doi: 10.1200/JCO.2012.47.7521. Epub 2013 Sep 16. No abstract available. PMID 24043743
- [Background] Besser MJ, Shapira-Frommer R, Itzhaki O, Treves AJ, Zippel DB, Levy D, Kubi A, Shoshani N, Zikich D, Ohayon Y, Ohayon D, Shalmon B, Markel G, Yerushalmi R, Apter S, Ben-Nun A, Ben-Ami E, Shimoni A, Nagler A, Schachter J. Adoptive transfer of tumor-infiltrating lymphocytes in patients with metastatic melanoma: intent-to-treat analysis and efficacy after failure to prior immunotherapies. Clin Cancer Res. 2013 Sep 1;19(17):4792-800. doi: 10.1158/1078-0432.CCR-13-0380. Epub 2013 May 20. PMID 23690483
- [Background] Pilon-Thomas S, Kuhn L, Ellwanger S, Janssen W, Royster E, Marzban S, Kudchadkar R, Zager J, Gibney G, Sondak VK, Weber J, Mule JJ, Sarnaik AA. Efficacy of adoptive cell transfer of tumor-infiltrating lymphocytes after lymphopenia induction for metastatic melanoma. J Immunother. 2012 Oct;35(8):615-20. doi: 10.1097/CJI.0b013e31826e8f5f. PMID 22996367
- [Background] Yeh S, Karne NK, Kerkar SP, Heller CK, Palmer DC, Johnson LA, Li Z, Bishop RJ, Wong WT, Sherry RM, Yang JC, Dudley ME, Restifo NP, Rosenberg SA, Nussenblatt RB. Ocular and systemic autoimmunity after successful tumor-infiltrating lymphocyte immunotherapy for recurrent, metastatic melanoma. Ophthalmology. 2009 May;116(5):981-989.e1. doi: 10.1016/j.ophtha.2008.12.004. PMID 19410956
- [Background] Johnson LA, Morgan RA, Dudley ME, Cassard L, Yang JC, Hughes MS, Kammula US, Royal RE, Sherry RM, Wunderlich JR, Lee CC, Restifo NP, Schwarz SL, Cogdill AP, Bishop RJ, Kim H, Brewer CC, Rudy SF, VanWaes C, Davis JL, Mathur A, Ripley RT, Nathan DA, Laurencot CM, Rosenberg SA. Gene therapy with human and mouse T-cell receptors mediates cancer regression and targets normal tissues expressing cognate antigen. Blood. 2009 Jul 16;114(3):535-46. doi: 10.1182/blood-2009-03-211714. Epub 2009 May 18. PMID 19451549
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- [Background] Malouf MA, Chhajed PN, Hopkins P, Plit M, Turner J, Glanville AR. Anti-viral prophylaxis reduces the incidence of lymphoproliferative disease in lung transplant recipients. J Heart Lung Transplant. 2002 May;21(5):547-54. doi: 10.1016/s1053-2498(01)00407-7. PMID 11983544